CLINICAL TRIAL: NCT03144505
Title: A 12-Month Randomized Control Trial in Patients With Type 2 Diabetes: Comparing Moderate and High-intensity Interval Training Protocols on Biomarkers and Quality of Life
Brief Title: Comparing Moderate and High-intensity Interval Training Protocols on Biomarkers in Type 2 Diabetes Patients
Acronym: D2FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: Associação Protectora dos Diabéticos de Portugal (Unknown)
Responsible Party: Principal Investigator, Luís Bettencourt Sardinha, Professor, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SFRH/BD/85742/2012
Record Dates: First submitted 2017-04-28; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Exercise; High Intensity Interval Training; Glycemic Control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): The control group will be invited to an orientation session, where it will be provided detailed information concerning their home base exercise program. Additionally, once in every 4 weeks, the control group will meet for thematic sessions regarding diabetes topics, such as, nutrition, physical activity, and clinical complications. Due to ethical reasons, the control group needs to be provided with a standard counseling approach, as suggested in this research project.
- MCT combined with RT Group (Experimental): MCT Group is designed to have equal energy expenditure when compared with HIIT Group. We standardized the exercise prescription according to body weight (kg), predicting that physical activity guidelines of 150 min peer week moderate intensity is equivalent to 10 kcal/kg of a combined session of RT and MCT. The MCT group will perform continuous cycling 3 days per week, with an exercise intensity of 40 to 59% of the heart rate reserve (HRR).
  Participants will also perform an RT circuit: 1 set of two pull upper body exercises (seated row and lat pulldown); 1 set of two push upper body exercises (chest press and shoulder press); 1 set of two leg exercises (leg press and one leg lunge); and 1 set of two core exercises (dead bug and regular plank). Each set consisting in 10 to 12 repetitions.
  Interventions: Behavioral: MCT combined with RT Group
- HIIT combined with RT Group (Experimental): The HIIT program will perform cycle ergometer 3 days a week, and it will be divided into three phases: preparation phase (weeks 1-4), where the participants perform MCT (40-59% of the HRR); transition phase (weeks 5-8), in which the HIIT program is introduced progressively, starting with bouts of 2 minutes at 70% of the HRR, followed by 1 minute at 40-59% of the HRR (weeks 5-6), and finishing with bouts of 80% of the HRR, followed by 1 minute at 40-59% of the HRR (weeks 7-8); training phase (weeks 9-42), where the participants perform 1 minute of exercise at 90% of the HRR, followed by 1 minute resting at 40-59% of the HRR.
  The HIIT session will have the same energy expenditure as the MCT group, using the 10kcal/kg week target. Participants will also fulfill the same RT as the MCT group.
  Interventions: Behavioral: HIIT combined with RT Group

INTERVENTIONS:
Behavioral: MCT combined with RT Group
  Arms: MCT combined with RT Group
Behavioral: HIIT combined with RT Group
  Arms: HIIT combined with RT Group

SUMMARY:
To overcome the lack of knowledge regarding the relative role of different intensities of aerobic training in adults with type 2 (T2D) diabetes, a 12 month randomized controlled trial will be performed to assess and compare the impact of two exercise groups: 1- high intensity interval training (HIIT) with resistance training; 2- moderate continuous training (MCT) with resistance training; and 3- a standard counseling home based control group; on hemoglobin A1c (HbA1c) as the main outcome, and other selected cardiometabolic, body composition and quality of life markers, as secondary outcomes. This investigation aims to increase the current knowledge on HIIT and the related benefits on diabetes control and treatment in a time saving and physiological efficient framework, which will improve the general health and well-being of the diabetes population. A total of 105 participants with T2D will be recruited from the Lisbon area (35 control, 35 HIIT, and 35 MCT). The investigators hypothesize that high-intensity interval training, compared to moderate continuous training, will optimize the physiological adaptations and quality of life in people with type 2 diabetes.

DETAILED DESCRIPTION:
Contemporary exercise guidelines focus on continuous aerobic exercise using mainly moderate intensity exercises. However, there is growing evidence that HIIT has the same (or even further) benefits, with lower time commitment. This type of exercise has already been tested in T2D patients, using mostly short intervention studies, with significant improvements in relevant outcomes for T2D, such as glucose regulation. On the other hand, no study as yet compared the effects of HIIT and MCT (both combining resistance training, RT) in a long-term study design. Therefore, this study will use a 12 month randomized control trial to assess the effects of an HIIT combined with RT, and MCT combined with RT, in comparison with a control group (home base program), on glycemic control, inflammatory profile, endothelium function, cardiorespiratory fitness, quality of life, and body composition outcomes, in adult males and females with T2D.

The sample recruitment is planned to be made using media, mails, and community events. Participants can be considered eligible if age is set between 30 and 75 years old, a body mass index lower than 48 kg/m2, and if they have been diagnosed with T2D (according to the ADA criteria). Further criteria will be made upon their medical history concerning strokes, advanced neuropathy or retinopathy, and other health conditions that may interfere with this study's protocols or otherwise safe exercising. Power and sample size calculations (G-Power, Version 3.1.3) are based on a predicted hemoglobinA1c difference of 0.66 hemoglobinA1c units with an SD of effect of 1.2 hemoglobinA1c units, α=0.05, 1-β=0.80 and an expected dropout rate of 10%. The calculations yielded a minimum sample size of 105 participants (35 in each group).

The statistical analysis will be performed using SPSS Statistics (version 22.0, SPSS Inc., an IBM Company, Chicago IL, USA). Baseline differences between the interventions and the control group will be examined using ANOVA, or a non-parametric alternative in case of a non-normalized distribution. Outcome variables will be analyzed using three-way mixed factorial ANOVA. Intention-to-treat analysis will be performed. Simple and multiple regression analysis will be performed to test the relationships among the selected variables. Statistical significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with type 2 diabetes
* 30-75 years of age
* BMI < 48 kg/m2

Exclusion Criteria:

* Documented cardiovascular disease
* Advanced neuropathy or retinopathy
* Physical health condition that may interfere with study's protocols or exercising safety

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Changes from baseline HbA1c at 3, 6, 9 and 12 months | 12 months
  Blood samples will be collected from an indwelling catheter for the assessment of HbA1c. Samples will be drawn into chilled, heparinized tubes and centrifuged rapidly to avoid glycolysis. HbA1c will be analyzed by immunoassay (auto analyzer Hb9210 Premier A. Menarini diagnostics).

SECONDARY OUTCOMES:
Changes from baseline cardiorespiratory fitness at 12 months | 12 months
  A stress test with ECG and gas analysis will be performed to assess cardiorepiratory fitness and to screen for eventual heart problems, under the supervision of appropriately trained medical staff.
Changes from baseline body composition at 3, 6, 9 and 12 months | 12 months
  Subjects weight and height will be measured according to standardized procedures. Waist circumference measurements will be done according to the NIH and WHO protocol. To estimate total and intra-abdominal fat mass and fat-free mass, DXA measurements will be made using a total body scan (Hologic Explorer-W, Waltham, USA).
Changes from baseline inflammatory profile at 12 months | 12 months
  This analysis will be done in standard inflammatory variables such as TNFα, PCR, IL-6 and cortisol.
Changes from baseline arterial function at 12 months | 12 months
  Arterial function assessment will be performed on the right carotid artery using an ultrasound scanner (MyLab One, Esaote, Genova, Italy) and implemented with a previously validated radiofrequency-based tracking of the arterial wall.
Changes from baseline quality of Life at 12 months | 12 months
  Quality of life will be measured using the SF-36 Health Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Luís Sardinha, Professor, Study Director — Professor

REFERENCES:
- [Derived] Correia IR, Hetherington-Rauth M, Magalhaes JP, Judice PB, Rosa GB, Henriques-Neto D, Manas A, Ara I, Silva AM, Sardinha LB. Compensatory mechanisms from different exercise intensities in type 2 diabetes: a secondary analysis of a 1-year randomized controlled trial. Acta Diabetol. 2023 May;60(5):645-654. doi: 10.1007/s00592-023-02038-7. Epub 2023 Feb 2. PMID 36729308
- [Derived] Magalhaes JP, Hetherington-Rauth M, Judice PB, Correia IR, Rosa GB, Henriques-Neto D, Melo X, Silva AM, Sardinha LB. Interindividual Variability in Fat Mass Response to a 1-Year Randomized Controlled Trial With Different Exercise Intensities in Type 2 Diabetes: Implications on Glycemic Control and Vascular Function. Front Physiol. 2021 Sep 16;12:698971. doi: 10.3389/fphys.2021.698971. eCollection 2021. PMID 34603073
- [Derived] Judice PB, Magalhaes JP, Hetherington-Rauth M, Correia IR, Sardinha LB. Sedentary patterns are associated with BDNF in patients with type 2 diabetes mellitus. Eur J Appl Physiol. 2021 Mar;121(3):871-879. doi: 10.1007/s00421-020-04568-2. Epub 2021 Jan 2. PMID 33389140
- [Derived] Magalhaes JP, Santos DA, Correia IR, Hetherington-Rauth M, Ribeiro R, Raposo JF, Matos A, Bicho MD, Sardinha LB. Impact of combined training with different exercise intensities on inflammatory and lipid markers in type 2 diabetes: a secondary analysis from a 1-year randomized controlled trial. Cardiovasc Diabetol. 2020 Oct 7;19(1):169. doi: 10.1186/s12933-020-01136-y. PMID 33028418
- [Derived] Hetherington-Rauth M, Magalhaes JP, Judice PB, Melo X, Sardinha LB. Vascular improvements in individuals with type 2 diabetes following a 1 year randomised controlled exercise intervention, irrespective of changes in cardiorespiratory fitness. Diabetologia. 2020 Apr;63(4):722-732. doi: 10.1007/s00125-020-05089-5. Epub 2020 Jan 20. PMID 31960071
- [Derived] Magalhaes JP, Melo X, Correia IR, Ribeiro RT, Raposo J, Dores H, Bicho M, Sardinha LB. Effects of combined training with different intensities on vascular health in patients with type 2 diabetes: a 1-year randomized controlled trial. Cardiovasc Diabetol. 2019 Mar 18;18(1):34. doi: 10.1186/s12933-019-0840-2. PMID 30885194